CLINICAL TRIAL: NCT00752180
Title: A Single Dose,Single Centre,Double Blind,Crossover Study Comparing the Pharmacokinetic Profiles of Wockhardt's Insulin Human Injection, Soluble (Recombinant DNA Origin) for Injection and Actrapid in Type 1 Diabetics
Brief Title: Comparative Glucose Clamp Study of Wockhardt's Insulin Human Regular for Injection and Actrapid, in Type 1 Diabetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wockhardt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: WosulinR/PK-PD/type1/EMEA/2008
Record Dates: First submitted 2008-09-12; First posted 2008-09-15 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-12

CONDITIONS: Diabetes
Keywords: pharmacokinetics; pharmacodynamics; type 1 diabetics; recombinant human insulin
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wosulin R (Experimental): Wosulin R,Regular insulin for injection(Recombinant Human Insulin)(600 nmol/ml, 100IU/ml)in vials 10.0 ml given subcutaneously.
  Interventions: Biological: Wosulin R
- Actrapid (Active Comparator): Actrapid, Regular insulin for injection (Recombinant Human Insulin) (600nmol/ml,100IU/ml)in vials 10.0 ml given subcutaneously.
  Interventions: Biological: Actrapid

INTERVENTIONS:
Biological: Wosulin R — Total dose per subject will be 0.3 IU/Kg given Subcutaneously.
  Arms: Wosulin R
Biological: Actrapid — Total dose per subject will be 0.3 IU/kg given Subcutaneously.
  Arms: Actrapid

SUMMARY:
The aim of this trial is to demonstrate bioequivalence of Wosulin R to Actrapid with regard to its total and to its maximum serum insulin concentrations.

DETAILED DESCRIPTION:
The purpose of this study is to test for bioequivalence based on the pharmacokinetic parameters Cmax and AUC0-12h between two recombinant soluble human insulin preparations. The study also compares the other pharmacokinetic parameters and pharmacodynamic profiles as well as assesses safety and local tolerability of the two insulin preparations in type 1 diabetics.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with type 1 diabetes mellitus
* Age between 18 and 45 years (both inclusive)
* Insulin treatment for at least 12 months before the screening visit
* Daily basal insulin requirement between 0.2 and 0.6 IU/kg/day (both inclusive) and current total daily insulin dose less than 1.2 IU/kg/day.
* Body Mass Index (BMI) between 18.0 and 35.0 kg/m2
* HbA1c less than or equal to 10.0%
* Fasting C-peptide < 0.4 nmol/L
* Non-smoker, no nicotine consumption for at least one year.
* Subjects considered generally healthy, except for the underlying diabetes mellitus and related morbidity (such as well controlled hypertension and dyslipidemia)
* Signed and dated informed consent obtained before any trial-related activities

Exclusion Criteria:

* Previous participation in this trial or other clinical trials within 30 days of dosing or 5 half-lives of any investigational drug, whichever is longer. If half life of the investigational drug is unknown, previous participation in other clinical trials within 3 months of dosing.
* Pregnant, breast-feeding or intention of becoming pregnant or not using adequate contraceptive measures (defined as intrauterine device that has been in place for at least 3 months, double barrier contraception, sterilization or abstinence, or oral contraceptive pill, which should have been taken without difficulty for at least 3 months, or an approved hormonal implant).
* Clinically significant abnormal hematology or biochemistry screening tests, as judged by the Investigator. In particular, subjects with elevated liver enzymes (AST or ALT > 2 times the upper limit of normal) or impaired renal function will not be allowed to enter the trial.
* Any serious systemic infectious disease during the four weeks prior to first dose of test drug,
* History of any illness that, in the opinion of the Investigator, might confound the results of the trial or pose risk in administering the trial drug to the subject. In particular, subjects with significant cardiovascular disease, anemia or hemoglobinopathy will not be allowed to enter the trial.
* Cardiac problems defined as: decompensated heart failure (NYHA class III and IV) at any time and/or angina pectoris and/or myocardial infarction within the last 12 months.
* Uncontrolled hypertension
* Subjects who have at screening, after 5 minutes rest, a supine blood pressure outside the range of 90-140 mmHg systolic or 50-90 mmHg diastolic, or pulse rate outside the range 40 to 90 beats per minute, or who are requiring more than two anti-hypertensive medications.
* Severe neuropathy (in particular autonomic neuropathy), retinopathy or maculopathy
* Clinically significant abnormal ECG at screening
* Recurrent major hypoglycemia or hypoglycemic unawareness as judged by the investigator or hospitalization for diabetic ketoacidosis during the 6 months preceding the screening visit.
* History of alcohol or drug abuse in the past five years and/or any positive test for drugs of abuse at screening.
* Positive test for hepatitis B or C or HIV
* Any systemic treatment with drugs known to interfere with glucose metabolism such as systemic corticoids, non-selective beta-blockers, thyroid hormone and monoamine oxidase inhibitors within 3 months prior to the first dosing visit.
* Use of drugs which may interfere with the interpretation of trial results or are known to cause clinically relevant interference with insulin action, glucose utilization or recovery from hypoglycemia
* Blood donation of more than 500 mL within the last 12 weeks
* History of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reaction
* Known or suspected allergy to trial products or related products
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or co-operation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2008-08; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Mean AUCins.0-12h and Cins.max | Visit 2 and 3

SECONDARY OUTCOMES:
PK endpoints: AUC0-4h, AUC0-6h, AUC6-12h,tmax, t½ and elimination rate constant.PD endpoints: AUCGIR0-4h, AUCGIR0-6h, AUCGIR6-12h, AUCGIR0-12h, GIRmax and tGIRmax .Safety endpoints: AEs, hematology, biochemistry, urinalyses, physical exam | Visit 2, 3 and 4

CONTACTS AND LOCATIONS:
Overall Officials: Till Schroer, Study Director — Profil Institute for Clinical Research, Inc.
Locations (1):
- Profil Institute for Clinical Research, Chula Vista, California, United States